CLINICAL TRIAL: NCT01447888
Title: Perioperative Pain Management In Spine Surgery Patients: Part I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3436-3
Record Dates: First submitted 2011-09-22; First posted 2011-10-06 (Estimated); Results first posted 2020-04-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Pain
Keywords: Spine surgery; Chronic pain; Opioid tolerant; Pain management in spine surgery patients
MeSH Terms: conditions — Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 150% Oral Morphine Equivalent (OME) (Experimental): Perioperative goal-directed opioid dosing at 150% of patient baseline oral morphine equivalent (OME) for opioid-tolerant patients
  Interventions: Drug: 150% Oral Morphine Equivalent (OME)
- Control (Active Comparator): Standard perioperative dosing, which does not currently account for patients' baseline opiate use.
  Interventions: Other: Clinical Judgment

INTERVENTIONS:
Drug: 150% Oral Morphine Equivalent (OME) — Patients will receive 150% of their oral morphine equivalent (OME) utilizing the drugs Dilaudid and Fentanyl.
  Arms: 150% Oral Morphine Equivalent (OME)
Other: Clinical Judgment — This method of perioperative parenteral opioid dosing has been used on spine surgery patients, based on clinical decision of the anesthesiologist.
  Arms: Control

SUMMARY:
The purpose of this study is a comparison of pain management in opioid-tolerant spine surgery patients using a perioperative dosing goal of 150% of patient's baseline oral morphine equivalent (OME), as compared to standard perioperative dosing, which does not currently account for patients' baseline opiate use.

DETAILED DESCRIPTION:
Spine surgery patients experience high levels of pain and report poor pain management in patient satisfaction surveys. Data examined from Allina HCAHPS (Hospital Consumer Assessment of Healthcare Providers and Systems) pain management questions indicate that spine surgery patients report poor pain management. In July, August, and September 2010 patients on the Abbott Northwestern (ANW) spine surgery unit reported 62% on the composite pain score compared to 69% to 71% for ANW overall. During these same three months, the proportion of patients on this unit reporting their pain was always well controlled ranged from 49% to 57% compared to 59% to 64% for the hospital overall. Since ANW serves a high number of spine surgery patients, this poor pain management reporting is a concern for patient care and possibly for future Medicare/Medicaid funding formulas.

Opioid-tolerant patients pose a particular challenge to pain management. The intervention to be tested specifically targets patients who are determined to be opioid-tolerant patients. Opioid-tolerant patients are generally patients who have severe chronic pain, and, thus, are taking pain medication regularly. Tolerance occurs when chronic exposure to a drug diminishes its analgesic effect or creates the need for a higher dose to maintain this effect. Given the severe chronic pain conditions of many patients who are presenting for spine surgery, there is a high level of opioid tolerance among these patients.

While there is no agreed upon definition in the literature about a fixed opioid amount that constitutes "opioid tolerance," Abbott Northwestern Hospital has a working definition of opioid tolerant patients as those who are receiving ≥ 20 mg of oxycodone (or equivalent)/day for > 7 days. This definition is slightly more aggressive than the Institute of Safe Medication Practices definition which set the standard at "at least 30 mg oxycodone/day for greater than a week."

While higher postoperative pain status has been documented in opioid-tolerant patients, very little has been done to examine customizing perioperative opioid dosing to improve pain management in this population. The proposed intervention is designed specifically to test if post-operative pain management can be improved in opioid-tolerant patients using perioperative goal-directed parenteral opioid dosing based on 150% of the patient's baseline oral morphine equivalent (OME). It is important to note this method of perioperative goal-directed parenteral opioid dosing has been used at ANW on spine surgery patients, based on clinical decision of the anesthesiologist. However, this strategy has not been tested compared to standard care.

For this study our research questions are:

1. Does the intervention improve immediate (4 hours) post-operative pain over the comparison group?
2. Does the intervention improve management during the 24 hours (or at discharge) after the recovery period over the comparison group?
3. Is the clinical intervention associated with selected improved post-operative status measures compared to the control group?
4. Is the clinical intervention associated with long-term differences in reported pain scores or medication levels as measured by a phone call at 4 weeks after surgery?

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years or older.
2. Patients must be undergoing spine surgery at ANW.
3. Patients must be assessed to be opioid tolerant based on the established criteria.
4. Patients must be willing and able to provide written informed consent.

Exclusion Criteria:

1. Patients unwilling to comply with research procedures.
2. Patients having surgery for correction of scoliosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-09; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Mrachek, MD, Principal Investigator — Allina Health System
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 150% Oral Morphine Equivalent (OME) | Control
Started | 45 | 55
Completed | 45 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 150% Oral Morphine Equivalent (OME) | Control | Total
Number analyzed (Participants) | 45 | 55 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (11.7) | 52 (12.6) | 51.55 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 32 | 47
  Male | 30 | 23 | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 45 | 55 | 100

OUTCOME MEASURES:

1. Primary Outcome: Immediate Postoperative Pain Control
Description: We will be assessing if the intervention improves immediate (4 hours) postoperative pain control as compared to the non-intervention group. Measures that will be used to assess immediate post-operative pain include: Verbal pain scores, opioid consumption, and vital signs. Verbal pain scores were reported using the Wong-Baker FACES pain rating scale which ranges from 0 (no hurt) to 10 (hurts worst). Higher numerical scores on the scale indicate more pain, thus a worse outcome.
Time Frame: 4 hours post surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 150% Oral Morphine Equivalent (OME) | Control
Number analyzed (Participants) | 45 | 55
score on a scale | 6.6 (2.1) | 6.8 (1.5)

2. Secondary Outcome: Pain Management Improvement at 24 Hours After the Recovery Period
Description: We will be assessing if the intervention improved postoperative pain management during the first 24 hours after the recovery period (first 4 hours postoperatively) as compared to the non-intervention group. Measures that will be used to assess success: Verbal pain scores, opioid consumption (doses and frequency), and vital signs. Verbal pain scores were reported using the Wong-Baker FACES pain rating scale which ranges from 0 (no hurt) to 10 (hurts worst). Higher numerical scores on the scale indicate more pain, thus a worse outcome.
Time Frame: 24 hours after the recovery period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 150% Oral Morphine Equivalent (OME) | Control
Number analyzed (Participants) | 45 | 55
score on a scale | 5.8 (2.0) | 6.4 (1.6)

ADVERSE EVENTS:
Time Frame: 24 hours post surgery
Description: Safety events to be examined in this research question include incidence of aspirations, emergent intubations, oxygen desaturation events, falls, hallucinations and/or delusions, and medication errors.
Arm/Group | 150% Oral Morphine Equivalent (OME) | Control
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/55
Other Adverse Events (participants affected / at risk) | 0/45 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No